CLINICAL TRIAL: NCT01860651
Title: Patient Empowerment: Web-based Monitoring in Children and Adolescents With Inflammatory Bowel Disease for Better Quality of Treatment
Brief Title: Web-based Monitoring in Children and Adolescents With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Katrine Carlsen, MD, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YOUNG-WEB
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-08

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn´s Disease
Keywords: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn´s Disease; Children; Adolescence; E-health web-monitoring; Adherence; Disease activity; Fecal Calprotectin
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Web-monitoring (Active Comparator): There is two arms for intervention:
  1) Patients in treatment with medicine administrated at home and 2) patients in treatment with biologicals.
  Interventions: Behavioral: Web-monitoring
- Control (No Intervention): Patients in treatment with medicine administrated at home: routine outpatient controls, four times a year.
  Patients in treatment with biologicals: retrospective routine treatment algorithm

INTERVENTIONS:
Behavioral: Web-monitoring — During the E-health intervention, symptoms and FC are monitored closely through the web-program and treatment will be initiated by symptoms and elevated FC.
  Arms: Web-monitoring

SUMMARY:
The investigators hypothesize that E-health - web based monitoring of disease and treatment - in young patients with chronic inflammatory disease (IBD) can improve the disease course and quality of life.

Adherence (to take the prescribed medicine) is difficult for young patients. In this E-health project the investigators seek to improve young patients (10-17 years) responsibility for treatment, to empower them and thereby enhance the adherence in order to achieve a more quiet disease course. Through the e-Health program and web-app the disease activity will be presented to the young patient via a simple traffic light chart and the patient will be guided to: continue the prescribed medication, call the physician or visit the out-patient clinic. In future the concept is believed also to be applicable for young patients with other chronic diseases.

DETAILED DESCRIPTION:
IBD's natural history is characterized by relapses (e.g. rectal bleeding, diarrhoea, abdominal pain, faecal urgency, fistula and anal abscess) and remissions. In children and adolescents the disease has a more aggressive course as compared with adults, causing a deterioration in the quality of life. During puberty patients are in an especially vulnerable period of their lives and there is a high risk for developing social disabilities due to the disease. Furthermore, IBD can lead to many days of absence from school and patients are at risk of not being able to maintain their education.

Patients are treated medically when the disease is active, but also in quiet phases too in order to maintain remission. It is therefore crucial for success that patients receive insight into the disease and understand the importance of following the recommended maintenance treatment. Despite being aware of an increased risk of acute hospitalization and surgery, it is difficult for both adult and pediatric patients to follow the continuous medication (adherence). It is known that up to 50% of young patients fail to take their medication as directed.

Previous studies have used E-health in the treatment of IBD patient. In M. Elkjaer et al. 2010 study on 300 patients with mild-to-moderate UC, E-health treatment resulted in shorter periods of active disease (average 18 vs. 77 days in the control group), 88% were satisfied with their treatment using E-health and the need for outpatient visits was reduced. In another study, Pedersen et al. 2012, on 27 patients with CD and examining biological treatment, E-Health was able to optimize the timing of infliximab treatment in CD patients. The E-Health solution was safe to use and patients showed high adherence to the program (86%). To the investigators knowledge no study has previously used E-health treatment in children and adolescents with IBD. It is, however, the investigators belief that this treatment concept would be readily taken up such patients, for whom web communication, at least in Denmark, is already a well-integrated part of their daily lives.

The current study consists of two projects: Project A: Patients in treatment with medicine administrated at home. Project B: Patients in treatment with biological infusions

Project A: Patients in treatment with medicine administrated at home are monitored, according to current international guidelines, with outpatient visits every third month. Patients participating in the current project will be randomly split into two groups and followed for two years. E-health group: Web-monitoring with an annual visit to the IBD center. Control group: Routine outpatient controls, four times a year.

Project B: According to current guidelines, patients receiving treatment with biologicals visit the outpatient clinic approximately every eighth week and treatment is given intravenously. During the E-health intervention, symptoms and fecal calprotectin are monitored closely through the web-program, and treatment will be initiated by symptoms and elevated FC. In this way the timing of treatment with biologicals can be optimized and infusions delayed with a maximum treatment-free period of 12 weeks, or earlier than 8 weeks if necessary.

ELIGIBILITY:
Inclusion Criteria:

* IBD diagnosis according to the Copenhagen and Porto criteria
* Aged between 10-17 years
* Fluent in Danish
* Access to the internet
* Patients in treatment with infliximab must have completed the induction period (i.e. minimum six week after start-up of treatment).

Exclusion Criteria:

* Insufficient Danish language skills
* Lack of intellectual capacity
* Growth retardation

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2013-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Carlsen, MD, Principal Investigator — Department of Pediatrics, Hvidovre Hospital; Vibeke Wewer, MD, PhD, Study Chair — Department of Pediatrics, Hvidovre Hospital; Pia Munkholm, Professor, Study Chair — Department of Gastroenterology, Herlev Hospital; Christian Jakobsen, MD, PhD, Study Chair — Department of Pediatrics, Hvidovre Hospital; Lene Riis, MD, PhD, Study Chair — Department of Pathology, Herlev Hospital
Locations (1):
- Department of Pediatrics, Hvidovre Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Carlsen K, Jakobsen C, Kallemose T, Paerregaard A, Riis LB, Munkholm P, Wewer V. F-calprotectin and Blood Markers Correlate to Quality of Life in Pediatric Inflammatory Bowel Disease. J Pediatr Gastroenterol Nutr. 2017 Nov;65(5):539-545. doi: 10.1097/MPG.0000000000001540. PMID 28169974

RESULTS

PARTICIPANT FLOW:
Groups:
- Web-monitoring: There is two arms for intervention:
  1) Patients in treatment with medicine administrated at home and 2) patients in treatment with biologicals.
  Web-monitoring: During the E-health intervention, symptoms and FC are monitored closely through the web-program and treatment will be initiated by symptoms and elevated FC.
- Control: Patients in treatment with medicine administrated at home: routine outpatient controls, four times a year.
  Patients in treatment with biologicals: routine treatment algorithm
Period: Overall Study
Arm/Group | Web-monitoring | Control
Started | 56 | 47
Completed | 31 | 39
Not Completed | 25 | 8

BASELINE CHARACTERISTICS:
Groups:
- Web-monitoring: There is two arms for intervention:
  Study 1) Patients in treatment with medicine administrated at home and Study 2) patients in treatment with biologicals.
- Control: Study 1) Patients in treatment with medicine administrated at home: routine outpatient controls, four times a year.
  Study 2) Patients in treatment with biologicals: retrospective routine treatment algorithm
- Total: Total of all reporting groups
Arm/Group | Web-monitoring | Control | Total
Number analyzed (Participants) | 56 | 47 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56 | 47 | 103
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.82) | 14.7 (2.11) | 14.9 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 22 | 53
  Male | 25 | 25 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 56 | 47 | 103
Region of Enrollment [Number; unit: participants]
  Denmark | 56 | 47 | 103

OUTCOME MEASURES:

1. Primary Outcome: Medical Adherence
Description: Participants (group 1, medication adm. at home): Medicine Adherence Report Scale (MARS): range 5-25 points. Higher scores mean a better outcome. In the below Outcome Measure Data Table the mean data for each group (web and control) summarized from the whole study periode are presented.
Time Frame: Prospective, each third month, up to 2 years
Population: Number of participants is only from study 1) Patients in treatment with medicine adminstered at home (participant in the web-group: 27; participant in the control-group: 26)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Web-monitoring: Patients in treatment with medicine administrated at home
  Web-monitoring: During the E-health intervention, symptoms and FC are monitored closely through the web-program and treatment will be initiated by symptoms and elevated FC.
- Control: Patients in treatment with medicine administrated at home: routine outpatient controls, four times a year.
Arm/Group | Web-monitoring | Control
Number analyzed (Participants) | 27 | 26
units on a scale | 23.3 [22.9 to 23.6] | 23.3 [22.9 to 23.7]
Statistical Analysis 1: Comparison: Web-monitoring vs Control; Statistical analysis of "Medical adherence" in study "Medication adm. at home" were analysed using a Mixed Effect Model (MEM). The MEM model included a random patient effect and a fixed effect interaction between group and time, to evaluate difference between the groups over time; Test type: Other; p = 0.22, Mixed Effect Model; mean difference over time = -0.002, 95% CI 2-sided [-0.005 to 0.001]

2. Secondary Outcome: Number of Participants With Step up in Medical Intensity
Description: Time to frist step-up in treatment intensity (escalating dose or change/addition of a more potent drug) were obtained from the patient's medical record during the study period, as a proxy of progression in disease activity.
  Time to step up was analysed via Kaplan Meier survival analysis.
Time Frame: The first event during participation (2 years). (events were prospecitvely registered)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Web-monitoring
Number analyzed (Participants) | 26 | 27
Participants | 10 | 12

3. Secondary Outcome: Surgery
Description: Need for surgery
Time Frame: The first event during participation (2 years). (events were prospecitvely registered)
Population: In this analysis both participants from study 1 (web 27, control 26) and 2 (web 29, control 21) are represented.
  No surgeries were performed, and therefore there is no mean and SD
Measure: Mean (Standard Deviation); unit: Surgeries
Arm/Group | Web-monitoring | Control
Number analyzed (Participants) | 56 | 47
Surgeries | 0 (0) | 0 (0)

4. Secondary Outcome: Absence From School
Description: Number of days absence from school
Time Frame: Prospective, each third month, - disease activity each month(project A) or week(project B), in 2 years
Measure: Mean (Standard Error); unit: days
Arm/Group | Web-monitoring | Control
Number analyzed (Participants) | 27 | 26
days | 1.6 (0.5) | 16.5 (4.4)

5. Secondary Outcome: Contact to the Hospital
Description: Need for outpatient visits
Time Frame: Prospective, each third month, - disease activity each month(project A) or week(project B), in 2 years
Measure: Median (Inter-Quartile Range); unit: visits
Arm/Group | Web-monitoring | Control
Number analyzed (Participants) | 27 | 26
visits | 2 [2 to 3] | 8 [4 to 9]

6. Secondary Outcome: Number of Weeks Between Treatment
Description: Date of IFX infusions were prospectively registered from both the eHealth and the control groups.
Time Frame: Prospective, each third month, - disease activity each month(project A) or week(project B), in 2 years
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Web-monitoring: Patients in treatment with biologicals.
- Control: Patients in treatment with biologicals: retrospective routine treatment algorithm
Arm/Group | Web-monitoring | Control
Number analyzed (Participants) | 29 | 21
weeks | 9.5 (2.3) | 6.9 (1.4)

ADVERSE EVENTS:
Time Frame: 2 ½ year
Description: Adverse Event that occured was allergic reactions during Infliximab infusions.
  Infusion related reactions was not collected in the biological control group. The control group was collected only to compare blood trough levels of IFX antibodies, IFX concentration, and treatment intervals. Therefore the total number of participants in the Adverse event tables representing participants in study 2 (patients in treatment with biologicals), only represents participants in the web-group.
Arm/Group | Web-monitoring | Control
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/26
Other Adverse Events (participants affected / at risk) | 3/29 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Web-monitoring (N=56) | Control (N=26)
Serious adverse event (Immune system disorders) | 0/27 (0) | 0 (0) — Data represents study 1. Description: events that would result in death, life-threatening events, prolongation of hospitalization or required intervention to prevent permanent impairment.
serious adverse events (Immune system disorders) | 0/29 (0) | 0/0 (0) — Data represents study 2. Serious event-data was not collected in the control group. Description: events that would result in death, life-threatening events, prolongation of hospitalization or required intervention to prevent permanent impairment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Web-monitoring (N=29) | Control (N=0)
Infusion-related allergic reactions (Immune system disorders) | 3 (3) | 0 (0) — Infliximab infusion-related allergic reactions was only collected in the web group in study 2 (Patients in treatment with biologicals). Data regarding infusion-related allergic reactions was not collected in the control group in study 2.

LIMITATIONS AND CAVEATS:
The main limitation is the relatively few participants that were all sourced from one center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-06-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT01860651/Prot_SAP_ICF_000.pdf